CLINICAL TRIAL: NCT02715726
Title: A Randomized, Double-blind, Parallel Group Study to Evaluate the Efficacy and Safety of Alirocumab (SAR236553/REGN727) Versus Ezetimibe in Asia in High Cardiovascular Risk Patients With Hypercholesterolemia Not Adequately Controlled With Their Statin Therapy
Brief Title: Evaluation of Alirocumab Versus Ezetimibe on Top of Statin in Asia in High Cardiovascular Risk Patients With Hypercholesterolemia
Acronym: ODYSSEY EAST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC13889; U1111-1150-8859 (Other: UTN)
Record Dates: First submitted 2016-03-16; First posted 2016-03-22 (Estimated); Results first posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab; Ezetimibe; Atorvastatin; Rosuvastatin Calcium; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ezetimibe 10 mg (Active Comparator): Oral ezetimibe 10 mg capsule once daily with or without food for 24 weeks and subcutaneous placebo injection for alirocumab every 2 weeks (Q2W) for 22 weeks added to lipid modifying therapy (LMT).
  Interventions: Drug: Placebo for alirocumab; Drug: ezetimibe; Drug: atorvastatin; Drug: rosuvastatin; Drug: simvastatin
- Alirocumab 75 mg Q2W/up to 150 mg Q2W (Experimental): Subcutaneous injection of alirocumab 75 mg Q2W and oral placebo capsule for ezetimibe once daily with or without food added to stable LMT for 24 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when LDL-C level was >=70 milligrams per deciliter (mg/dL) (1.81 millimoles per liter [mmol/L]) at Week 8.
  Interventions: Drug: Alirocumab; Drug: placebo for ezetimibe; Drug: atorvastatin; Drug: rosuvastatin; Drug: simvastatin

INTERVENTIONS:
Drug: Alirocumab — Pharmaceutical form:solution Route of administration: subcutaneous
  Other Names: SAR236553 (REGN727)
  Arms: Alirocumab 75 mg Q2W/up to 150 mg Q2W
Drug: Placebo for alirocumab — Pharmaceutical form:solution Route of administration: subcutaneous
  Arms: Ezetimibe 10 mg
Drug: ezetimibe — Pharmaceutical form:capsule Route of administration: oral
  Arms: Ezetimibe 10 mg
Drug: placebo for ezetimibe — Pharmaceutical form:capsule Route of administration: oral
  Arms: Alirocumab 75 mg Q2W/up to 150 mg Q2W
Drug: atorvastatin — Pharmaceutical form:tablet Route of administration: oral
Drug: rosuvastatin — Pharmaceutical form:tablet Route of administration: oral
Drug: simvastatin — Pharmaceutical form:tablet Route of administration: oral

SUMMARY:
Primary Objective:

To demonstrate the reduction of low-density lipoprotein cholesterol (LDL-C) by alirocumab as add-on therapy to stable maximally tolerated daily statin therapy in comparison to ezetimibe 10 mg daily after 24 weeks of treatment in Asia in participants with hypercholesterolemia at high cardiovascular (CV) risk.

Secondary Objectives:

* To evaluate the effect of alirocumab 75 mg in comparison with ezetimibe 10 mg on LDL-C after 12 weeks of treatment.
* To evaluate the effect of alirocumab on other lipid parameters: e.g., apolipoprotein B (Apo B), non-high density lipoprotein cholesterol (non-HDL-C), total cholesterol (TC), lipoprotein a (Lp[a]), HDL-C, triglycerides (TG), apolipoprotein A-1 (Apo A-1).
* To evaluate the safety and tolerability of alirocumab.
* To evaluate the development of anti-alirocumab antibodies.
* To evaluate the pharmacokinetics (PK) of alirocumab.

DETAILED DESCRIPTION:
The maximum study duration was 35 weeks per participant, which included a screening period of up to 3 weeks, a 24-week randomized treatment period, and an 8-week post-treatment follow-up period.

ELIGIBILITY:
Inclusion criteria:

Participants with hypercholesterolemia and established coronary heart disease (CHD) or CHD risk equivalents who are not adequately controlled with a maximally tolerated daily dose of statin at a stable dose for at least 4 weeks prior to the screening visit (Week -3).

Exclusion criteria:

* Participants without established CHD or CHD risk equivalents.
* LDL-C <70 mg/dL (<1.81 mmol/L) at the screening visit (Week -3) in participants with history of documented CV disease.
* LDL-C <100 mg/dL (<2.59 mmol/L) at the screening visit (Week -3) in participants without history of documented CV disease.
* Change in statin dose or dose regimen from screening to randomization.
* Currently taking a statin other than atorvastatin, rosuvastatin, or simvastatin.
* Atorvastatin, rosuvastatin, or simvastatin was not taken daily or not taken at a registered dose.
* Daily doses above atorvastatin 80 mg, rosuvastatin 40 mg, or simvastatin 40 mg.
* Use of cholesterol absorption inhibitor (ie, ezetimibe), omega-3 fatty acid (at doses ≥1000 mg daily), nicotinic acid, fibrates, bile acid-binding sequestrant, or red yeast rice products in the past 4 weeks prior to screening visit (Week -3).
* Fasting serum triglycerides >400 mg/dL (>4.52 mmol/L) at the screening period.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 615 (Actual)
Dates: Start 2016-07-27 (Actual); Primary Completion 2018-08-06 (Actual); Study Completion 2018-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (62):
- China (41):
  - Investigational Site Number 1560027, Beijing
  - Investigational Site Number 1560043, Beijing
  - Investigational Site Number 1560039, Beijing
  - Investigational Site Number 1560012, Beijing
  - Investigational Site Number 1560018, Beijing
  - Investigational Site Number 1560006, Changchun
  - Investigational Site Number 1560020, Changchun
  - Investigational Site Number 1560023, Changsha
  - Investigational Site Number 1560030, Fuzhou
  - Investigational Site Number 1560005, Guangzhou
  - Investigational Site Number 1560040, Guangzhou
  - Investigational Site Number 1560025, Guangzhou
  - Investigational Site Number 1560048, Hangzhou
  - Investigational Site Number 1560037, Hangzhou
  - Investigational Site Number 1560008, Hangzhou
  - Investigational Site Number 1560014, Hohhot
  - Investigational Site Number 1560016, Jinan
  - Investigational Site Number 1560044, Lanzhou
  - Investigational Site Number 1560028, Nanchang
  - Investigational Site Number 1560045, Nanjing
  - Investigational Site Number 1560017, Nanjing
  - Investigational Site Number 1560031, Nanjing
  - Investigational Site Number 1560035, Nanning
  - Investigational Site Number 1560029, Shanghai
  - Investigational Site Number 1560041, Shanghai
  - Investigational Site Number 1560053, Shanghai
  - Investigational Site Number 1560009, Shenyang
  - Investigational Site Number 1560001, Shenyang
  - Investigational Site Number 1560042, Shenyang
  - Investigational Site Number 1560036, Shenzhen
  - Investigational Site Number 1560056, Siping
  - Investigational Site Number 1560021, Taiyuan
  - Investigational Site Number 1560002, Tianjin
  - Investigational Site Number 1560022, Tianjin
  - Investigational Site Number 1560052, Tianjin
  - Investigational Site Number 1560055, Wenzhou
  - Investigational Site Number 1560003, Wuhan
  - Investigational Site Number 1560004, Xi'an
  - Investigational Site Number 1560019, Xuzhou
  - Investigational Site Number 1560054, Yinchuan
  - Investigational Site Number 1560057, Zhanjiang
- India (17):
  - Investigational Site Number 3560017, Belagavi
  - Investigational Site Number 3560001, Gūrgaon
  - Investigational Site Number 3560003, Hubli
  - Investigational Site Number 3560010, Kolkata
  - Investigational Site Number 3560019, Kolkata
  - Investigational Site Number 3560020, Mangalore
  - Investigational Site Number 3560006, Mumbai
  - Investigational Site Number 3560007, Nagpur
  - Investigational Site Number 3560004, Nagpur
  - Investigational Site Number 3560008, Nagpur
  - Investigational Site Number 3560016, Nagpur
  - Investigational Site Number 3560014, New Delhi
  - Investigational Site Number 3560005, Pune
  - Investigational Site Number 3560011, Pune
  - Investigational Site Number 3560013, Surat
  - Investigational Site Number 3560015, Vijayawada
  - Investigational Site Number 3560012, Vijaywada
- Thailand (4):
  - Investigational Site Number 7640004, Bangkok
  - Investigational Site Number 7640003, Bangkok Noi
  - Investigational Site Number 7640001, Muang
  - Investigational Site Number 7640002, Pratumwan

REFERENCES:
- [Derived] Han Y, Chen J, Chopra VK, Zhang S, Su G, Ma C, Huang Z, Ma Y, Yao Z, Yuan Z, Zhao Q, Kuanprasert S, Baccara-Dinet MT, Manvelian G, Li J, Chen R. ODYSSEY EAST: Alirocumab efficacy and safety vs ezetimibe in high cardiovascular risk patients with hypercholesterolemia and on maximally tolerated statin in China, India, and Thailand. J Clin Lipidol. 2020 Jan-Feb;14(1):98-108.e8. doi: 10.1016/j.jacl.2019.10.015. Epub 2019 Nov 18. PMID 31882376

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 61 centers in China, India and Thailand. Overall 1163 participants were screened between 27 July 2016 and 18 December 2017, of whom 548 were screen failures. Screen failures were mainly due to exclusion criteria met. A total of 615 participants were randomized in 2:1 ratio to alirocumab: ezetimibe.
Pre-assignment Details: Randomization was stratified according to prior history of myocardial infarction (MI) or ischemic stroke [Yes/No], and high-intensity statin treatment (Yes: atorvastatin 40 to 80 mg daily or rosuvastatin 20 to 40 mg daily, no: atorvastatin below 40 mg daily, rosuvastatin below 20 mg daily or simvastatin whatever the dose daily) and country.
Groups:
- Alirocumab 75 mg Q2W/up to 150 mg Q2W: Subcutaneous injection of alirocumab 75 mg Q2W and oral placebo capsule for ezetimibe once daily with or without food added to stable LMT for 24 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when low-density lipoprotein cholesterol (LDL-C) level was >=70 milligrams per deciliter (mg/dL) (1.81 millimoles per liter [mmol/L]) at Week 8.
Period: Overall Study
Arm/Group | Ezetimibe 10 mg | Alirocumab 75 mg Q2W/up to 150 mg Q2W
Started | 208 (Randomized) | 407 (Randomized)
Treated | 207 | 405
Safety Population (1 participant of ezetimibe arm received alirocumab: counted in alirocumab arm for safety analysis.) | 206 | 406
Completed | 190 | 380
Not Completed | 18 | 27
Not completed — Adverse Event | 2 | 6
Not completed — Protocol Violation | 1 | 0
Not completed — Death | 2 | 1
Not completed — Participant moved | 1 | 3
Not completed — Other than specified above | 11 | 15
Not completed — Randomized but not treated | 1 | 2

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized participants.
Groups:
- Ezetimibe 10 mg: Oral ezetimibe 10 mg capsule once daily with or without food for 24 weeks and subcutaneous placebo injection for alirocumab Q2W for 22 weeks added to LMT.
- Alirocumab 75 mg Q2W/up to 150 mg Q2W: Subcutaneous injection of alirocumab 75 mg Q2W and oral placebo capsule for ezetimibe once daily with or without food added to stable LMT for 24 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when LDL-C level was >=70 mg/dL (1.81 mmol/L) at Week 8.
- Total: Total of all reporting groups
Arm/Group | Ezetimibe 10 mg | Alirocumab 75 mg Q2W/up to 150 mg Q2W | Total
Number analyzed (Participants) | 208 | 407 | 615
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.3 (11.2) | 58.8 (10.7) | 58.6 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 92 | 154
  Male | 146 | 315 | 461
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 208 | 407 | 615
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Calculated LDL-C in mmol/L [Mean (Standard Deviation); unit: mmol/L] — Calculated LDL-C in mmol/L from Friedewald formula (LDL-C = Total cholesterol - High-density lipoprotein cholesterol [HDL-C] - [Triglyceride/2.2]).
  mmol/L | 2.875 (1.287) | 2.862 (1.253) | 2.866 (1.264)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Calculated Low Density Lipoprotein Cholesterol at Week 24: Intent-to-treat (ITT) Analysis
Description: Adjusted least square (LS) means and standard errors at Week 24 were obtained from mixed models analysis with repeated measures (MMRM) to account for missing data. All available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment were used in the model (ITT analysis).
Time Frame: From Baseline to Week 24
Population: ITT population included all randomized participants with one baseline and at least one post-baseline calculated LDL-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75 mg Q2W/up to 150 mg Q2W
Number analyzed (Participants) | 208 | 403
percent change | -20.3 (2.0) | -56.0 (1.5)
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Alirocumab 75 mg Q2W/up to 150 mg Q2W; Alirocumab group was compared to ezetimibe group using an appropriate contrast statement; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS mean difference = -35.6, 95% CI 2-sided [-40.6 to -30.7] — Alirocumab 75 mg Q2W/up to 150 mg Q2W vs. Ezetimibe

2. Secondary Outcome: Percent Change From Baseline in Calculated Low Density Lipoprotein Cholesterol at Week 24: On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 24 were obtained from MMRM model including all available post-baseline on-treatment data from Week 4 to Week 24 (i.e. up to 21 days after last injection or 3 days after the last capsule, whichever came first) (on-treatment analysis).
Time Frame: From Baseline to Week 24
Population: Modified ITT (mITT) population included all randomized and treated participants with one baseline and at least one post-baseline calculated LDL-C value on-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75 mg Q2W/up to 150 mg Q2W
Number analyzed (Participants) | 204 | 401
percent change | -21.3 (2.0) | -58.7 (1.4)
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Alirocumab 75 mg Q2W/up to 150 mg Q2W; A hierarchical testing method was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when previous endpoint was statistically significant at 0.05 level; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS mean difference = -37.3, 95% CI 2-sided [-42.1 to -32.6] — Alirocumab 75 mg Q2W/up to 150 mg Q2W vs. Ezetimibe

3. Secondary Outcome: Percent Change From Baseline in Calculated Low Density Lipoprotein Cholesterol at Week 12: ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 were obtained from MMRM model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 12
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75 mg Q2W/up to 150 mg Q2W
Number analyzed (Participants) | 208 | 403
percent change | -22.2 (1.9) | -57.1 (1.4)
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Alirocumab 75 mg Q2W/up to 150 mg Q2W; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant); Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS mean difference = -34.9, 95% CI 2-sided [-39.5 to -30.2] — Alirocumab 75 mg Q2W/up to 150 mg Q2W vs. Ezetimibe

4. Secondary Outcome: Percent Change From Baseline in Calculated Low Density Lipoprotein Cholesterol at Week 12: On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 12 were obtained from MMRM model including all available post-baseline on-treatment data from Week 4 to Week 24 (i.e. up to 21 days after last injection or 3 days after the last capsule, whichever came first) (on-treatment analysis).
Time Frame: From Baseline to Week 12
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75 mg Q2W/up to 150 mg Q2W
Number analyzed (Participants) | 204 | 401
percent change | -22.7 (1.9) | -58.1 (1.4)
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Alirocumab 75 mg Q2W/up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS mean difference = -35.4, 95% CI 2-sided [-40.0 to -30.7] — Alirocumab 75 mg Q2W/up to 150 mg Q2W vs. Ezetimibe

5. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (Apo B) at Week 24: ITT Analysis
Description: Adjusted LS means and standard errors at Week 24 were obtained from MMRM model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline Apo B value on- or off-treatment (Apo B ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent Change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75 mg Q2W/up to 150 mg Q2W
Number analyzed (Participants) | 203 | 398
percent Change | -16.2 (1.4) | -43.5 (1.0)
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Alirocumab 75 mg Q2W/up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — Threshold for significance at 0.05 level; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS mean difference = -27.4, 95% CI 2-sided [-30.8 to -23.9] — Alirocumab 75 mg Q2W/up to 150 mg Q2W vs. Ezetimibe

6. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at Week 24: On-Treatment Analysis
Description: as for outcome 2
Time Frame: From Baseline to Week 24
Population: Participants of the mITT population with one baseline and at least one post-baseline Apo B value on-treatment (Apo B mITT population).
Measure: Least Squares Mean (Standard Error); unit: percent Change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75 mg Q2W/up to 150 mg Q2W
Number analyzed (Participants) | 197 | 392
percent Change | -17.4 (1.4) | -45.2 (1.0)
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Alirocumab 75 mg Q2W/up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS mean difference = -27.8, 95% CI 2-sided [-31.2 to -24.4] — Alirocumab 75 mg Q2W/up to 150 mg Q2W vs. Ezetimibe

7. Secondary Outcome: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol (Non-HDL-C) at Week 24: ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline non-HDL-C value on- or off-treatment (non-HDL-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent Change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75 mg Q2W/up to 150 mg Q2W
Number analyzed (Participants) | 208 | 403
percent Change | -19.4 (1.7) | -47.0 (1.2)
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Alirocumab 75 mg Q2W/up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS mean difference = -27.7, 95% CI 2-sided [-31.8 to -23.6] — Alirocumab 75 mg Q2W/up to 150 mg Q2W vs. Ezetimibe

8. Secondary Outcome: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol at Week 24: On-Treatment Analysis
Description: as for outcome 2
Time Frame: From Baseline to Week 24
Population: Participants of the mITT population with one baseline and at least one post-baseline non-HDL-C value on-treatment (non-HDL-C mITT population).
Measure: Least Squares Mean (Standard Error); unit: percent Change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75 mg Q2W/up to 150 mg Q2W
Number analyzed (Participants) | 204 | 401
percent Change | -20.4 (1.7) | -49.1 (1.2)
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Alirocumab 75 mg Q2W/up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS mean difference = -28.7, 95% CI 2-sided [-32.6 to -24.7] — Alirocumab 75 mg Q2W/up to 150 mg Q2W vs. Ezetimibe

9. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (Total-C) at Week 24: ITT Analysis
Description: Adjusted LS means and standard errors at Week 24 were obtained from MMRM model including all available post-baseline data from Week 4 up to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: Participants from the ITT population with one baseline and at least one post-baseline Total-C value on- or off-treatment (Total-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent Change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75 mg Q2W/up to 150 mg Q2W
Number analyzed (Participants) | 208 | 403
percent Change | -13.8 (1.2) | -33.9 (0.9)
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Alirocumab 75 mg Q2W/up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS mean difference = -20.2, 95% CI 2-sided [-23.1 to -17.2] — Alirocumab 75 mg Q2W/up to 150 mg Q2W vs. Ezetimibe

10. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at Week 12: ITT Analysis
Description: as for outcome 3
Time Frame: From Baseline to Week 12
Population: Apo B ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent Change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75 mg Q2W/up to 150 mg Q2W
Number analyzed (Participants) | 203 | 398
percent Change | -16.5 (1.4) | -43.0 (1.0)
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Alirocumab 75 mg Q2W/up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS mean difference = -26.5, 95% CI 2-sided [-29.8 to -23.2] — Alirocumab 75 mg Q2W/up to 150 mg Q2W vs. Ezetimibe

11. Secondary Outcome: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol at Week 12: ITT Analysis
Description: as for outcome 3
Time Frame: From Baseline to Week 12
Population: Non-HDL-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent Change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75 mg Q2W/up to 150 mg Q2W
Number analyzed (Participants) | 208 | 403
percent Change | -20.7 (1.6) | -47.4 (1.1)
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Alirocumab 75 mg Q2W/up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS mean difference = -26.7, 95% CI 2-sided [-30.5 to -22.8] — Alirocumab 75 mg Q2W/up to 150 mg Q2W vs. Ezetimibe

12. Secondary Outcome: Percent Change From Baseline in Total Cholesterol at Week 12: ITT Analysis
Description: as for outcome 3
Time Frame: From Baseline to Week 12
Population: Total-C ITT population
Measure: Least Squares Mean (Standard Error); unit: percent Change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75 mg Q2W/up to 150 mg Q2W
Number analyzed (Participants) | 208 | 403
percent Change | -14.9 (1.2) | -34.2 (0.8)
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Alirocumab 75 mg Q2W/up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS mean difference = -19.3, 95% CI 2-sided [-22.1 to -16.5] — Alirocumab 75 mg Q2W/up to 150 mg Q2W vs. Ezetimibe

13. Secondary Outcome: Percentage of Participants Reaching Calculated Low Density Lipoprotein Cholesterol <70 mg/dL (1.81 mmol/L) at Week 24: ITT Analysis
Description: Adjusted percentages at Week 24 were obtained from multiple imputation approach for handling of missing data. All available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment were included in the imputation model.
Time Frame: Up to Week 24
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Ezetimibe 10 mg | Alirocumab 75 mg Q2W/up to 150 mg Q2W
Number analyzed (Participants) | 208 | 403
percentage of participants | 40.5 | 85.1
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Alirocumab 75 mg Q2W/up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — Threshold for significance at 0.05 level; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 11.2, 95% CI 2-sided [7.1 to 17.7] — Alirocumab 75 mg Q2W/up to 150 mg Q2W vs Ezetimibe

14. Secondary Outcome: Percentage of Participants Reaching Calculated Low Density Lipoprotein Cholesterol <70 mg/dL (1.81 mmol/L) at Week 24: On-Treatment Analysis
Description: Adjusted percentages at Week 24 were obtained from multiple imputation approach including all available post-baseline on-treatment data from Week 4 to Week 24 (i.e. up to 21 days after last injection or 3 days after the last capsule, whichever came first) (on-treatment analysis).
Time Frame: Up to Week 24
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Ezetimibe 10 mg | Alirocumab 75 mg Q2W/up to 150 mg Q2W
Number analyzed (Participants) | 204 | 401
percentage of participants | 42.1 | 87.0
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Alirocumab 75 mg Q2W/up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — Threshold for significance at 0.05 level; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 13.6, 95% CI 2-sided [8.3 to 22.3] — Alirocumab 75 mg Q2W/up to 150 mg Q2W vs Ezetimibe

15. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) (Lp[a]) at Week 24: ITT Analysis
Description: Adjusted means and standard errors at Week 24 were obtained from multiple imputation approach followed by robust regression model for handling missing data. All available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment were included in the imputation model.
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Mean (Standard Error); unit: percent Change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75 mg Q2W/up to 150 mg Q2W
Number analyzed (Participants) | 208 | 403
percent Change | 3.956 (2.095) | -30.317 (1.461)
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Alirocumab 75 mg Q2W/up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Robust — Threshold for significance at 0.05 level; Multiple imputation approach followed by a robust regression model; Adjusted Mean Difference = -34.273, 95% CI 2-sided [-39.262 to -29.285] — Alirocumab 75 mg Q2W/up to 150 mg Q2W vs. Ezetimibe

16. Secondary Outcome: Percent Change From Baseline in High Density Lipoprotein Cholesterol at Week 24: ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline HDL-C value on- or off-treatment (HDL-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75 mg Q2W/up to 150 mg Q2W
Number analyzed (Participants) | 208 | 403
percent change | 6.5 (1.3) | 8.3 (0.9)
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Alirocumab 75 mg Q2W/up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.2280, Mixed Models Analysis — Threshold for significance at 0.05 level; LS mean difference = 1.9, 95% CI 2-sided [-1.2 to 4.9] — Alirocumab 75 mg Q2W/up to 150 mg Q2W vs. Ezetimibe

17. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides (TG) at Week 24: ITT Analysis
Description: Adjusted means and standard errors at Week 24 were obtained by using multiple imputation approach followed by robust regression model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75 mg Q2W/up to 150 mg Q2W
Number analyzed (Participants) | 208 | 403
percent change | -14.409 (1.904) | -14.462 (1.341)

18. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A-1 (Apo A-1) at Week 24: ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 24
Population: Participants from the ITT population with one baseline and at least one post-baseline Apo A-1 value on- or off-treatment (Apo A-1 ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75 mg Q2W/up to 150 mg Q2W
Number analyzed (Participants) | 203 | 398
percent change | -0.2 (0.8) | 3.2 (0.6)

19. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) at Week 12: ITT Analysis
Description: Adjusted means and standard errors at Week 12 were obtained from multiple imputation approach followed by robust regression model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 12
Population: ITT population.
Measure: Mean (Standard Error); unit: percent Change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75 mg Q2W/up to 150 mg Q2W
Number analyzed (Participants) | 208 | 403
percent Change | 6.313 (2.056) | -30.064 (1.449)

20. Secondary Outcome: Percent Change From Baseline in High Density Lipoprotein Cholesterol at Week 12: ITT Analysis
Description: as for outcome 3
Time Frame: From Baseline to Week 12
Population: HDL-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75 mg Q2W/up to 150 mg Q2W
Number analyzed (Participants) | 208 | 403
percent change | 6.1 (1.2) | 7.3 (0.9)

21. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 12: ITT Analysis
Description: Adjusted means and standard errors at Week 12 were obtained by using multiple imputation approach followed by a robust regression model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 12
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75 mg Q2W/up to 150 mg Q2W
Number analyzed (Participants) | 208 | 403
percent change | -13.585 (1.929) | -9.965 (1.379)

22. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A-1 at Week 12 : ITT Analysis
Description: as for outcome 3
Time Frame: From Baseline to Week 12
Population: Apo A-1 ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75 mg Q2W/up to 150 mg Q2W
Number analyzed (Participants) | 203 | 398
percent change | 1.1 (0.8) | 3.7 (0.6)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to 32 weeks of the study regardless of seriousness or relationship to investigational product.
Description: Reported AEs were treatment emergent AEs that developed or worsened during 'the treatment emergent period' (time from first dose of double-blind study drug intake [capsule or injection, whichever came first] to the day of last dose of double blind study drug injection + 70 days). Analysis was performed on safety population (participants who received at least 1 dose or partial dose of study drug [injection or capsule)]. Participants were analyzed according to the treatment actually received.
Groups:
- Alirocumab 75 mg Q2W/up150 mg Q2W: Subcutaneous injection of alirocumab 75 mg Q2W and oral placebo capsule for ezetimibe once daily with or without food added to stable LMT for 24 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when LDL-C level was >=70 mg/dL (1.81 mmol/L) at Week 8.
Arm/Group | Ezetimibe 10 mg | Alirocumab 75 mg Q2W/up150 mg Q2W
All-Cause Mortality (participants affected / at risk) | 3/206 | 2/406
Serious Adverse Events (participants affected / at risk) | 23/206 | 41/406
Other Adverse Events (participants affected / at risk) | 41/206 | 71/406
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe 10 mg (N=206) | Alirocumab 75 mg Q2W/up150 mg Q2W (N=406)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 3 (3) | 3 (3)
Angina Unstable (Cardiac disorders) | 0 (0) | 9 (9)
Arrhythmia Supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 1 (1) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac Failure Acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 2 (3) | 0 (0)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Sudden Hearing Loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhagic Erosive Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Obstructive Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 2 (2) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0)
Anal Abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Lung Infection (Infections and infestations) | 1 (1) | 1 (1)
Necrotising Soft Tissue Infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 4 (5)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Brain Herniation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subarachnoid Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Limb Mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain Oedema (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral Arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral Artery Occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral Infarction (Nervous system disorders) | 0 (0) | 1 (2)
Cerebral Ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular Insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic Cerebral Infarction (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic Stroke (Nervous system disorders) | 2 (2) | 0 (0)
Loss Of Consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Adnexa Uteri Cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe 10 mg (N=206) | Alirocumab 75 mg Q2W/up150 mg Q2W (N=406)
Upper Respiratory Tract Infection (Infections and infestations) | 29 (39) | 54 (69)
Accidental Overdose (Injury, poisoning and procedural complications) | 15 (21) | 27 (40)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-10-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT02715726/SAP_000.pdf
  • Study Protocol (2015-12-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT02715726/Prot_001.pdf